CLINICAL TRIAL: NCT03812471
Title: Optimization of Fetal Biometry With 3D Ultrasound and Image Recognition
Acronym: EPICEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Electronics Nederland B.V. acting through Philips CTO organization (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ICBE-2-24301
Record Dates: First submitted 2018-09-06; First posted 2019-01-23 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Main study: 3D volumes acquisitions (Experimental): 3D volume acquisitions
  Interventions: Device: 3D volume acquisitions
- Ancillary study: 2D and 3D acquisitions (Experimental): 2D standard measurements and 3D volumes acquisitions
  Interventions: Device: 2D standard measurements and 3D volumes acquisitions

INTERVENTIONS:
Device: 3D volume acquisitions — 2 abdominal volumes 2 thigh volumes 2 head volumes
  Arms: Main study: 3D volumes acquisitions
Device: 2D standard measurements and 3D volumes acquisitions — * 1 abdomen circumference measurement
  * 1 femur length measurement
  * 1 head circumference measurement
  * 1 bi-parietal diameter measurement
  * 1 abdominal volume
  * 1 thigh volume
  * 1 head volume
  Arms: Ancillary study: 2D and 3D acquisitions

SUMMARY:
In the proposed clinical investigation, the investigational device (BabySize3D) will provide automated plane extraction and automated biometry measurements from 3D US volumes. The results obtained from the investigational software

ELIGIBILITY:
Inclusion Criteria:

* evolutive pregnancy with one fetus with a Gestational Age between 16 and 30 weeks
* aged between 18 and 65 years.
* social welfare benefit recipient
* willing and able to provide informed consent

Exclusion Criteria:

* under 18 years old
* multiple pregnancy
* over 18 years old and mentioned in French law articles L.1126-6 et L-1126-8,
* fetal malformation or suspected fetal malformation
* technical conditions that do not allow for standard fetal biometry (abdominal wall, fetal position, BMI > 25 kg/m2)
* fetal biometry non indicated in the standard pregnancy follow-up
* unwilling or unable to provide informed consent (e. g. physical, mental disability or linguistic factor that compromises patient information)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2023-03-17 (Actual)

PRIMARY OUTCOMES:
Bi-parietal diameter in mm. | Day 1
  The bi-parietal diameter in mm will be obtained with three methods: (1) fully automated 3D volume processing and caliper placement, (2) manual 3D volume processing and caliper placement, (3) manual selection of the 2D view plane and manual caliper placement on the screen of the ultrasound system (corresponding to standard of care measurements). The values obtained with the three methods and the differences between these values will be reported.
Head circumference in mm | Day 1
  The Head circumference in mm will be obtained with three methods: (1) fully automated 3D volume processing and caliper placement, (2) manual 3D volume processing and caliper placement, (3) manual selection of the 2D view plane and manual caliper placement on the screen of the ultrasound system (corresponding to standard of care measurements). The values obtained with the three methods and the differences between these values will be reported.
Abdominal circumference in mm | Day 1
  The Abdominal circumference in mm will be obtained with three methods: (1) fully automated 3D volume processing and caliper placement, (2) manual 3D volume processing and caliper placement, (3) manual selection of the 2D view plane and manual caliper placement on the screen of the ultrasound system (corresponding to standard of care measurements). The values obtained with the three methods and the differences between these values will be reported.
Femur length in mm | Day 1
  The Femur length in mm will be obtained with three methods: (1) fully automated 3D volume processing and caliper placement, (2) manual 3D volume processing and caliper placement, (3) manual selection of the 2D view plane and manual caliper placement on the screen of the ultrasound system (corresponding to standard of care measurements). The values obtained with the three methods and the differences between these values will be reported

SECONDARY OUTCOMES:
Failure rate of the automated measurements | Day 1
  Failure rate of the automated measurements
Exam and post-processing duration | Day 1
  Exam and post-processing duration
Difference of scores of the 2D standard cephalic plane and cephalic plane extracted from the 3D volume, based on six criteria listed in (Salomon et al. Ultrasound Obstet Gynecol 2006; 27: 34-40) | Day 1
  The cephalic plane extracted from the 3D volume and the 2D standard cephalic plane will be scored according to the six criteria described in (Salomon et al. Ultrasound Obstet Gynecol 2006; 27: 34-40). The scores and their difference will be reported.
Difference of scores of the 2D standard abdominal plane and abdominal plane extracted from the 3D volume, based on six criteria listed in (Salomon et al. Ultrasound Obstet Gynecol 2006; 27: 34-40) | Day 1
  The abdominal plane extracted from the 3D volume and the 2D standard abdominal plane will be scored according to the six criteria described in (Salomon et al. Ultrasound Obstet Gynecol 2006; 27: 34-40). The scores and their difference will be reported.
Difference of scores of the 2D standard femoral plane and femoral plane extracted from the 3D volume, based on four criteria listed in (Salomon et al. Ultrasound Obstet Gynecol 2006; 27: 34-40) | Day 1
  The femoral plane extracted from the 3D volume and the 2D standard femoral plane will be scored according to the four criteria described in (Salomon et al. Ultrasound Obstet Gynecol 2006; 27: 34-40). The scores and their difference will be reported.
Difference of scores of (i) the 2D standard cephalic plane and of (ii) the frames of a sequence of 2D images including the fetus head (cine-loop), based on six criteria listed in (Salomon et al. Ultrasound Obstet Gynecol 2006; 27: 34-40) | Day 1
  The 2D standard cephalic plane and the frames of a sequence of 2D images including the fetus head will be scored according to the six criteria described in (Salomon et al. Ultrasound Obstet Gynecol 2006; 27: 34-40). The scores and the score difference (standard view score - frame score) will be reported.
Difference of scores of (i) the 2D standard abdominal plane and of (ii) the frames of a sequence of 2D images including the fetus abdomen (cine-loop), based on six criteria listed in (Salomon et al. Ultrasound Obstet Gynecol 2006; 27: 34-40) | Day 1
  The 2D standard abdominal plane and the frames of a sequence of 2D images including the fetus abdomen will be scored according to the six criteria described in (Salomon et al. Ultrasound Obstet Gynecol 2006; 27: 34-40). The scores and the score difference (standard view score - frame score) will be reported.
Difference of scores of (i) the 2D standard femoral plane and of (ii) the frames of a sequence of 2D images including the fetus femur (cine-loop), based on four criteria listed in (Salomon et al. Ultrasound Obstet Gynecol 2006; 27: 34-40) | Day 1
  The 2D standard femoral plane and the frames of a sequence of 2D images including the fetus femur will be scored according to the four criteria described in (Salomon et al. Ultrasound Obstet Gynecol 2006; 27: 34-40). The scores and the score difference (standard view score - frame score) will be reported.
Title: Intraclass correlation coefficient of the bi-parietal diameter in mm (same operator) | Day 1
  The intraclass correlation coefficient of the bi-parietal diameter in mm measured from two different 3D volumetric acquisitions of the same patient performed by the same operator will be calculated.
Bland-Altman representation of the bi-parietal diameter in mm (same operator) | Day 1
  A Bland-Altman representation of the the bi-parietal diameter in mm measured from two different 3D volumetric acquisitions of the same patient performed by the same operator will be built.
Intraclass correlation coefficient of the bi-parietal diameter in mm (different operators) | Day 1
  The intraclass correlation coefficient of the bi-parietal diameter in mm measured from the 3D volumetric acquisitions of the same patient performed by two different operators will be calculated.
Bland-Altman representation of the bi-parietal diameter in mm (different operators) | Day 1
  A Bland-Altman representation of the bi-parietal diameter in mm measured from the 3D volumetric acquisitions of the same patient performed by two different operators will be built.
Intraclass correlation coefficient of the head circumference in mm (same operator) | Day 1
  the intraclass correlation coefficient of the head circumference in mm measured from two different 3D volumetric acquisitions of the same patient performed by the same operator will be calculated.
Bland-Altman representation of the head circumference in mm (same operator) | Day 1
  A Bland-Altman representation of the head circumference in mm measured from two different 3D volumetric acquisitions of the same patient performed by the same operator will be built.
Intraclass correlation coefficient of the head circumference in mm (different operators) | Day 1
  The intraclass correlation coefficient of the head circumference in mm measured from the 3D volumetric acquisitions of the same patient performed by two different operators will be calculated.
Bland-Altman representation of the head circumference in mm (different operators) | Day 1
  A Bland-Altman representation of the head circumference in mm measured from the 3D volumetric acquisitions of the same patient performed by two different operators will be built.
Intraclass correlation coefficient of the abdominal circumference in mm (same operator) | Day 1
  The intraclass correlation coefficient of the abdominal circumference in mm measured from two different 3D volumetric acquisitions of the same patient performed by the same operator will be calculated.
Bland-Altman representation of the abdominal circumference in mm (same operator) | Day 1
  A Bland-Altman representation of the abdominal circumference in mm measured from two different 3D volumetric acquisitions of the same patient performed by the same operator will be built.
Intraclass correlation coefficient of the abdominal circumference in mm (different operators) | Day 1
  The intraclass correlation coefficient of the abdominal circumference in mm measured from the 3D volumetric acquisitions of the same patient performed by two different operators will be calculated.
Bland-Altman representation of the abdominal circumference in mm (different operators) | Day 1
  A Bland-Altman representation of the abdominal circumference in mm measured from the 3D volumetric acquisitions of the same patient performed by two different operators built.
Intraclass correlation coefficient of the femoral length in mm (same operator) | Day 1
  The intraclass correlation coefficient of the femoral length in mm measured from two different 3D volumetric acquisitions of the same patient performed by the same operator will be calculated.
Bland-Altman representation of the femoral length in mm (same operator) | Day 1
  A Bland-Altman representation of the femoral length in mm measured from two different 3D volumetric acquisitions of the same patient performed by the same operator will be built.
Title: Intraclass correlation coefficient of the femoral length in mm (different operators) | Day 1
  The intraclass correlation coefficient of the femoral length in mm measured from the 3D volumetric acquisitions of the same patient performed by two different operators will be calculated.
Bland-Altman representation of the femoral length in mm (different operators) | Day 1
  A Bland-Altman representation of the femoral length in mm measured from the 3D volumetric acquisitions of the same patient performed by two different operators will be built.

CONTACTS AND LOCATIONS:
Overall Officials: Gaëlle Gaëlle AMBROISE-GRANDJEAN, Principal Investigator — CHRU de Nancy
Locations (1):
- CHRU de Nancy Brabois, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ambroise Grandjean G, Hossu G, Banasiak C, Ciofolo-Veit C, Raynaud C, Rouet L, Morel O, Beaumont M. Optimization of Fetal Biometry With 3D Ultrasound and Image Recognition (EPICEA): protocol for a prospective cross-sectional study. BMJ Open. 2019 Dec 15;9(12):e031777. doi: 10.1136/bmjopen-2019-031777. PMID 31843832